CLINICAL TRIAL: NCT06273657
Title: Effects of Medisinstart for Type 2 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Apokus AS (Other)
Collaborators: Norwegian Pharmacy Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Apokus-002
Record Dates: First submitted 2024-02-01; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Type 2 Diabetes
Keywords: Medication related problems; Adherence; Type 2 diabetes; Pharmacist-led intervention; Consultation; Pharmacy
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medisinstart (Experimental)
  Interventions: Other: Medisinstart
- Control (No Intervention)

INTERVENTIONS:
Other: Medisinstart — Medisinstart is a counseling service in pharmacies where patients who start taking a new medicine receive two follow-up consultations with a pharmacist.
  Arms: Medisinstart

SUMMARY:
Medisinstart is a counseling service in pharmacies where patients who start taking a new medicine receive two follow-up appointments with a pharmacist. The aim of the service is to promote correct medication use and increase patient adherence. The effect of Medisinstart has previously been studied among patients starting a new cardiovascular drug. The aim of the project is to map the effects of Medisinstart among patients starting a new medication for type 2 diabetes. Knowledge about the effects of Medisinstart is important in order to maximize the benefits of the service for patients and society. The project is being conducted as a randomized controlled trial among adult patients starting a new medication for type 2 diabetes. The intervention group receives Medisinstart, while the control group only receives prescription dispensing as normal. Data collection includes HbA1c analysis in blood samples and responses to questionnaires. HbA1c is an established measure of glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* Extracted a new drug/active substance (A10A/A10B) for type 2 diabetes
* Age ≥ 18 years
* The drugs are administered by the patient/relatives
* Good command of Norwegian, both written and spoken

Exclusion Criteria:

* Inability to understand and/or complete consent forms, questionnaires and/or other patient-oriented materials
* Not able to attend physical appointments in the pharmacy
* Not given written consent to participate in the study
* Diabetes medication is administered by a healthcare professional
* Known pregnancy
* HbA1c is unsuitable as an average measure of blood glucose at baseline
* Received initiation of medication for type 2 diabetes within the last year
* Ongoing participation in other studies involving similar interventions to increase adherence and ensure correct medication use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
HbA1c | At baseline and 6 months after initation of the new medication for type 2 diabetes.
  Change in HbA1c-level from baseline to 6 months after initiation of a new medication for type 2 diabetes.
HbA1c | At baseline and 12 months after initation of the new medication for type 2 diabetes.
  Change in HbA1c-level from baseline to 12 months after initiation of a new medication for type 2 diabetes.

SECONDARY OUTCOMES:
Self-reported adherence | 6 and 12 months after initiation of the new medication for type 2 diabetes
  Adherence will be measured by a Norwegian translation of the MARS-5 questionnaire. The total MARS-5 score can have values from 5-25, with higher scores indicating higher adherence.
Self-reported adherence | 6 and 12 months after initiation of the new medication for type 2 diabetes
  Adherence will be measured by a Norwegian translations of the question: "People often miss taking doses of their medicines, for a wide range of reasons. Have you missed any doses of your new medicine the last week?" The question will be answered by yes/no.
Frequency of medication-related problems | At the first and second Medisinstart consultations and 12 months after initiation of the new medication for type 2 diabetes
  Pharmacists will report identified medication-related problems (MRPs) in a structured self-developed electronic questionnaire. The MRP categories in the questionnaire are based on the MRP classification presented by Ruths et al. (Tidsskr Nor Laegeforen. 2007 Nov 29;127(23):3073-6). The different MRP categories will be reported as identified or not identified in the consultations.
Patients' beliefs about their medicines | At baseline and 6 months after initation of the new medication for type 2 diabetes
  Patients' beliefs about their medicines will be measured by a validated Norwegian translation of the Beliefs about Medicines Questionnaire (BMQ). The BMQ general comprises three subscales, Harm, Overuse and Benefit, and the total score of each subscale ranges from 4 to 20. The BMQ specific comprises two subscales, Concerns and Necessity, and the total score of each subscale ranges from 5 to 25. Higher scores indicate stronger beliefs in the concepts represented by the subscale.
Diabetes Self-Management | 12 months after initiation of the new medication for type 2 diabetes
  Diabetes Self-Management will be measured by a validated Norwegian translation of the Diabetes Self-Management Questionnaire-Revised (DSMQ-R). The scores are summed and transformed into a 1-10 scale for each of the following activities: "eating behavior", "medication use", "glucose monitoring", "physical activity" and "interaction with treating physician/healthcare professional". In addition, a total score is calculated as an overall measure of the patient's diabetes self-management. Values in the upper part of the scale indicate good self-care.
Diabetes Treatment Satisfaction | At baseline and 6 and 12 months after initiation of the new medication for type 2 diabetes
  Diabetes Treatment Satisfaction will be measured by a validated Norwegian translation of the Diabetes Treatment Satisfaction Questionnaire (DTSQ). The scores range from 0 to 36 where higher scores indicate greater satisfaction with treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Bremer, PhD, Principal Investigator — Head of Research and Development
Locations (19):
- Norway (19):
  - Ryfylke apotek, Rennesøy, Rennesøy
  - Apotek 1 Veakrossen, Veavåg, Veavåg
  - Vitusapotek Åfjord, Åfjord
  - Apotek 1 Andslimoen, Bardufoss
  - Apotek 1 Brandbu, Brandbu
  - Apotek 1 Brummundal, Brumunddal
  - Sykehusapoteket i Drammen, Drammen
  - Vitusapotek Gjøvik, Gjøvik
  - Vitusapotek Jessheim, Jessheim
  - Boots apotek Kløfta, Kløfta
  - Vitusapotek Leksvik, Leksvik
  - Apotek 1 Lena, Lena
  - Boots apotek Loddefjord, Loddefjord
  - Sykehusapoteket i Oslo, Aker, Oslo
  - Vitusapotek Røa, Oslo
  - Vitusapotek Jekta, Tromsø
  - Sykehusapoteket i Trondheim, Trondheim
  - Vitusapotek Ulefoss, Ulefoss
  - Boots apotek Linnea, Øystese

IPD SHARING:
Plan to Share IPD: No